CLINICAL TRIAL: NCT05792748
Title: A Clinical Trial Comparing Reinforced Zinc Oxide Eugenol to Ferric Sulphate as a Pulpotomy Agent in Primary Teeth
Brief Title: Comparison of Zinc Oxide Eugenol to Ferric Sulphate Pulpotomy in Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19/2013
Record Dates: First submitted 2023-02-24; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Pulpotomy
Keywords: Ferric sulphate; Zinc Oxide Eugenol; Pulpotomy; Primary dentition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZOE group (Active Comparator): Pulp hemostasis achieved by a dry cotton pellet applied on the pulp, then the chamber was filled with reinforced zinc oxide eugenol (ZOE) directly over the pulp.
  Interventions: Procedure: Pulp hemostasis with a dry cotton pellet; Procedure: Stainless steel crown
- FS group (Active Comparator): Pulp hemostasis achieved by a wet cotton pellet impregnated with ferric sulphate (FS) applied on the pulp, then the chamber was filled with (ZOE) directly over the pulp.
  Interventions: Procedure: Pulp hemostasis with a wet cotton pellet impregnated with FS; Procedure: Stainless steel crown

INTERVENTIONS:
Procedure: Pulp hemostasis with a dry cotton pellet — Application of a dry cotton pellet, then the chamber was filled with ZOE directly over the pulp
  Arms: ZOE group
Procedure: Pulp hemostasis with a wet cotton pellet impregnated with FS — Application of a a wet cotton pellet impregnated with FS, then the chamber was filled with ZOE directly over the pulp
  Arms: FS group
Procedure: Stainless steel crown — Stainless steel crown placed as a final restoration

SUMMARY:
In this prospective randomized, single blinded; split-mouth clinical trial the aim was to evaluate clinical and radiographic effects of placement of reinforced zinc oxide eugenol (ZOE) base directly over the amputated pulp stumps in pulpotomized primary molars, and to compare this technique to ferric sulphate (FS) in pulpotomized primary teeth. Included were 65 children using a split-mouth design, (130 teeth). All teeth were then restored with prefabricated stainless steel crowns (SSC). Patients were recalled for clinical and radiographical evaluation after 3, 6, 12 and 24 months. Two experienced and calibrated pediatric dentists who were not involved in the investigation blindly assessed the radiographs.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study was to evaluate the clinical and radiographic effects of placement of reinforced zinc oxide eugenol (ZOE) base directly over the amputated pulp stumps in pulpotomized primary molars, and to compare the effects of this technique to ferric sulphate (FS) agent in pulpotomized primary teeth.

Methods:

A sample of 65 children with bilateral deep carious mandibular primary molars who attended the pediatric dental clinics, at Jordan University of Science and Technology (JUST) were selected for this prospective randomized, single blinded; split-mouth clinical trial. The teeth were randomly divided into 2 treatment groups: in the ZOE group (n=65 teeth) hemostasis was achieved by a dry cotton pellet, then the chamber was filled with zinc oxide eugenol (ZOE) directly over the pulp on one side. In the FS group (n=65 teeth) hemostasis was achieved by a wet cotton pellet, ferric sulphate (FS) was applied on the pulp, then the chamber was filled with (ZOE) on the contralateral side. All teeth were restored with prefabricated stainless steel crowns (SSC). Patients were recalled for evaluation clinically after 1month, then clinically and radiographically after 3, 6, 12 and 24 months. Two experienced and calibrated pediatric dentists who were not involved in the investigation blindly assessed the radiographs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children
* Child has cooperative behaviour in the dental chair
* No history of spontaneous pain
* Deep caries in the tooth
* Carious exposure of a vital pulp
* A restorable tooth after completion of the pulp treatment
* Healthy periapical tissue on pre-operative periapical radiograph

Exclusion Criteria:

* Presence of tenderness to percussion and/or mobility
* Pathologic radiographic signs on pre-operative periapical radiograph including external or internal root resorption, calcification in the canal, periodontal membrane widening, periapical pathology, and furcation radiolucency.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2013-01-02 (Actual); Primary Completion 2014-01-02 (Actual); Study Completion 2014-04-01 (Actual)

PRIMARY OUTCOMES:
Number of teeth which are asymptomatic without clinical signs of disease | 24 months
  including percussion sensitivity, spontaneous pain, mobility, or abscess (Clinical)
Number of teeth with no pathological changes present | 24 months
  including radiolucency, root or bone resorption (Radiographic)

CONTACTS AND LOCATIONS:
Overall Officials: Ola B. Al-Batayneh, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Briso AL, Rahal V, Mestrener SR, Dezan Junior E. Biological response of pulps submitted to different capping materials. Braz Oral Res. 2006 Jul-Sep;20(3):219-25. doi: 10.1590/s1806-83242006000300007. PMID 17119704
- [Background] Casas MJ, Layug MA, Kenny DJ, Johnston DH, Judd PL. Two-year outcomes of primary molar ferric sulfate pulpotomy and root canal therapy. Pediatr Dent. 2003 Mar-Apr;25(2):97-102. PMID 12723832
- [Background] Casas MJ, Kenny DJ, Johnston DH, Judd PL. Long-term outcomes of primary molar ferric sulfate pulpotomy and root canal therapy. Pediatr Dent. 2004 Jan-Feb;26(1):44-8. PMID 15080357
- [Background] Chien MM, Setzer S, Cleaton-Jones P. How does zinc oxide-eugenol compare to ferric sulphate as a pulpotomy material? SADJ. 2001 Mar;56(3):130-5. PMID 16894712
- [Background] Fei AL, Udin RD, Johnson R. A clinical study of ferric sulfate as a pulpotomy agent in primary teeth. Pediatr Dent. 1991 Nov-Dec;13(6):327-32. PMID 1843987
- [Background] Hansen HP, Ravn JJ, Ulrich D. Vital pulpotomy in primary molars. A clinical and histologic investigation of the effect of zinc oxide-eugenol cement and Ledermix. Scand J Dent Res. 1971;79(1):13-25. No abstract available. PMID 5292960
- [Background] Hui-Derksen EK, Chen CF, Majewski R, Tootla RG, Boynton JR. Retrospective record review: reinforced zinc oxide-eugenol pulpotomy: a retrospective study. Pediatr Dent. 2013 Jan-Feb;35(1):43-6. PMID 23635897
- [Background] Huth KC, Paschos E, Hajek-Al-Khatar N, Hollweck R, Crispin A, Hickel R, Folwaczny M. Effectiveness of 4 pulpotomy techniques--randomized controlled trial. J Dent Res. 2005 Dec;84(12):1144-8. doi: 10.1177/154405910508401210. PMID 16304444
- [Background] Huth KC, Hajek-Al-Khatar N, Wolf P, Ilie N, Hickel R, Paschos E. Long-term effectiveness of four pulpotomy techniques: 3-year randomised controlled trial. Clin Oral Investig. 2012 Aug;16(4):1243-50. doi: 10.1007/s00784-011-0602-3. Epub 2011 Aug 13. PMID 21842145
- [Background] Ibricevic H, al-Jame Q. Ferric sulfate as pulpotomy agent in primary teeth: twenty month clinical follow-up. J Clin Pediatr Dent. 2000 Summer;24(4):269-72. doi: 10.17796/jcpd.24.4.d7u6405nw1132705. PMID 11314410
- [Background] Markovic D, Zivojinovic V, Vucetic M. Evaluation of three pulpotomy medicaments in primary teeth. Eur J Paediatr Dent. 2005 Sep;6(3):133-8. PMID 16216093
- [Background] Oliveira TM, Moretti AB, Sakai VT, Lourenco Neto N, Santos CF, Machado MA, Abdo RC. Clinical, radiographic and histologic analysis of the effects of pulp capping materials used in pulpotomies of human primary teeth. Eur Arch Paediatr Dent. 2013 Apr;14(2):65-71. doi: 10.1007/s40368-013-0015-x. Epub 2013 Apr 3. PMID 23549993
- [Background] Papagiannoulis L. Clinical studies on ferric sulphate as a pulpotomy medicament in primary teeth. Eur J Paediatr Dent. 2002 Sep;3(3):126-32. PMID 12871001
- [Background] Waterhouse PJ, Nunn JH, Whitworth JM, Soames JV. Primary molar pulp therapy--histological evaluation of failure. Int J Paediatr Dent. 2000 Dec;10(4):313-21. doi: 10.1046/j.1365-263x.2000.00211.x. PMID 11310245
- [Background] Zurn D, Seale NS. Light-cured calcium hydroxide vs formocresol in human primary molar pulpotomies: a randomized controlled trial. Pediatr Dent. 2008 Jan-Feb;30(1):34-41. PMID 18402097